CLINICAL TRIAL: NCT01423734
Title: Pilot Study To Assess The Reproducibility Of Diffusion Weighted Magnetic Resonance Imaging For Neuroendocrine Tumor Liver Metastases
Brief Title: The Reproducibility Of Diffusion Weighted Magnetic Resonance Imaging For Neuroendocrine Tumor Liver Metastases
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 11-122
Record Dates: First submitted 2011-08-24; First posted 2011-08-26 (Estimated); Last update posted 2023-01-23 (Actual); Status verified 2023-01

CONDITIONS: Gastro-enteropancreatic Neuroendocrine Tumor; Secondary Malignant Neoplasm of Liver
Keywords: ADRENAL GLAND; MRI; 11-122
MeSH Terms: conditions — Gastro-enteropancreatic neuroendocrine tumor | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- MRI: Patients will be consented for a second MRI without additional intravenous contrast, referred to from now on as 'research MRI', to be performed later on the same day as their clinical liver MR examination, on one of two 3.0 Tesla MR 750 GE scanners at the Breast and Imaging Center. The research MRI will consist only of the localizer and diffusion weighted imaging (DWI) sequences, with acquisition parameters identical to our clinical MRI. The reproducibility of DWI is best assessed in separate MR imaging sessions, although the examinations can be performed the same day.
  Interventions: Other: magnetic resonance imaging (MRI)

INTERVENTIONS:
Other: magnetic resonance imaging (MRI) — Each patient will undergo clinical and research MRI examinations. Before any MRI examination, the patient will answer a standard radiology MR department questionnaire form, with specific questions addressing contra-indications to MRI. The questionnaire form will be reviewed by radiology personnel as per standard practice.
  During the research MRI, the patient will be monitored visually and communication will be maintained between the patient and the MR technologists via a speaker system. At the termination of the study, the patient will be evaluated by the MR department radiology personnel as done routinely. Two breath hold DWI sequences will be performed for each patient. Since this is a reproducibility study, identical scan parameters will be used for the clinical and research MRI. The multiple b value DWI will be performed using the enhanced DW sequence that have been recently made available on our 3.0 Tesla MR 750 scanners at the Breast and Imaging Center.

SUMMARY:
Imaging with CT (Computed Tomography) or MRI (Magnetic Resonance Imaging) is normally used to see how tumors respond to treatment. If tumors shrink after therapy, doctors continue with the same treatment. On the other hand, growing tumors in a patient can bring about a change in therapy. Unfortunately, it often takes three to six months, or even longer before the investigators see tumors shrink or grow on scans. Doctors are looking for new imaging tools that can look at how tumors respond early on during treatment. This study will help us decide if such an MRI technology called DWI (Diffusion Weighted Imaging) can be used as a helpful imaging tool.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologic evidence of well differentiated neuroendocrine tumor of gastroenteropancreatic origin
* Evidence of metastatic disease of at least 2.0 cm in the liver by MRI or CT imaging.
* Patient ≥18 years of age on the day of signing informed consent.

Exclusion Criteria:

* Any contraindication to MRI based on departmental MR questionnaire
* Inability to cooperate for an MR exam
* Patient has a history of a second active malignancy with evidence of metastases. Patients with a history of resected prior malignancy or one that would not interfere with the MRI results is allowed.
* Patient has known psychiatric or substance abuse disorders that would, in the opinion of the treating investigator, interfere with cooperation with the requirements of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential research patients will be identified by doctors from the Gastrointestinal Oncology Service.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2011-08-23 (Actual); Primary Completion 2023-01-19 (Actual); Study Completion 2023-01-19 (Actual)

PRIMARY OUTCOMES:
reproducibility of diffusion weighted imaging for neuroendocrine liver metastases. | 2 years
  The investigators will calculate an ADC value for each metastasis that was chosen through consensus by the two participating radiologists. ADC is a voxel-level measurement so summary measures will be employed in order to get a single measurement for the ROI of each metastasis under study. For both the clinical and research MRI, the investigators will take the voxel-level data and calculate the mean, median, and minimum ADC within each ROI.

SECONDARY OUTCOMES:
evaluate the repeatability of perfusion insensitive diffusion coefficients ADC high of liver metastases | 2 years
  A similar application of the CCC will be employed to assess both intra-observer and interobserver variability separately for ADC high as in the primary aim. The repeatability and reproducibility of the ADC high will then be compared to the most repeatable and reproducible ADC measures identified in Aim 1 by ranking the CCC values and selecting the measure with the highest value.
evaluate the reproducibility perfusion insensitive diffusion coefficients (ADC high) of liver metastases | 2 years
  A similar application of the CCC will be employed to assess both intra-observer and interobserver variability separately for ADC high as in the primary aim. The repeatability and reproducibility of the ADC high will then be compared to the most repeatable and reproducible ADC measures identified in Aim 1 by ranking the CCC values and selecting the measure with the highest value.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Kinh Gian Do, MD,PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm